CLINICAL TRIAL: NCT04876157
Title: Artificial Intelligence-aimed Point-of-care Ultrasound Image Interpretation System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202006124RINC
Record Dates: First submitted 2021-05-02; First posted 2021-05-06 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Ultrasound Image Interpretation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Artificial intelligence-aimed ultrasound image interpretation (Experimental)
  Interventions: Diagnostic Test: Artificial intelligence-aimed point-of-care ultrasound image interpretation system

INTERVENTIONS:
Diagnostic Test: Artificial intelligence-aimed point-of-care ultrasound image interpretation system — improve the sensitivity and specificity of the AI-aimed ultrasound interpretation system

SUMMARY:
This proposal is for an one-year project. In this project, we aim to investigate the feasibility of using AI for sonographic image interpretation. The main project is responsible for coordination between the two sub-projects and the main project, providing image resources, and using U-Net (Convolutional Networks for Biomedical Image Segmentation) and Transfer Learning to build up the models for image recognition and validating the efficacy of the models. The purpose of Subproject 1 is to develop an image recognition system for dynamic images: pericardial effusion. After building up the model, validating the efficacy and future revision will be done. Subproject 2 comes out an image recognition system for static images: hydronephrosis. After building up the model, validating the efficacy and future revision will be done.

DETAILED DESCRIPTION:
Ultrasound is a non-invasive and non-radiated diagnostic tool in the emergency and critical care settings. In clinical practice, timely interpretation of sonographic images to facilitate decision-making is essential. However, it depends on operators' experience. As usual, it takes time for junior emergency physicians to have good diagnostic accuracy through traditional sonographic education. How to shorten the learning This proposal is for an one-year project. In this project, we aim to investigate the feasibility of using AI for sonographic image interpretation. The main project is responsible for coordination between the two sub-projects and the main project, providing image resources, and using U-Net (Convolutional Networks for Biomedical Image Segmentation) and Transfer Learning to build up the models for image recognition and validating the efficacy of the models. The purpose of Subproject 1 is to develop an image recognition system for dynamic images: pericardial effusion. After building up the model, validating the efficacy and future revision will be done. Subproject 2 comes out an image recognition system for static images: hydronephrosis. After building up the model, validating the efficacy and future revision will be done.

This pioneer study can provide two AI-assisted ultrasound image recognition systems in the real clinical conditions. They can experience of clinical applications and contribute to current medical education. Moreover, it can improve decision-making process and quality of care in the emergency and critical care units. Furthermore, the set-up models can be used in other target ultrasound image recognition in the future.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving echocardiography or renal ultrasound

Exclusion Criteria:

* patients not receiving echocardiography or renal ultrasound

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of AI interpretation | 6 months
  increase the sensitivity and specificity of AI to interpret the ultrasound image

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Wan-Ching Lien, Taipei, None Selected, Taiwan

IPD SHARING:
Plan to Share IPD: No